CLINICAL TRIAL: NCT00709722
Title: Safety and Efficacy Study on Deoxyspergualin (NKT-01) in Patients With Uncontrolled Lupus Nephritis Receiving Oral Corticosteroids and Prior Treatment of Standard Immunosuppressive Therapy
Brief Title: Safety and Efficacy on Deoxyspergualin (NKT-01) in Patients With Lupus Nephritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nippon Kayaku Co., Ltd. (Industry)
Responsible Party: Peter A. Heinzel, Ph.D., Clinical and Scientific Department, Euro Nippon Kayaku GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLE01-ENK
Record Dates: First submitted 2008-07-02; First posted 2008-07-03 (Estimated); Results first posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2008-07

CONDITIONS: Lupus Nephritis
Keywords: Lupus nephritis; Deoxyspergualin; Immunosuppression
MeSH Terms: conditions — Lupus Nephritis | interventions — gusperimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): NKT-01
  Interventions: Drug: NKT-01

INTERVENTIONS:
Drug: NKT-01 — SC, 0.5 mg/kg/day, consecutive 14 days administrations, 1 week rest, 9 cycles.
  Other Names: Deoxyspergualin, gusperimus

SUMMARY:
The aim of the open multi-center study is to determine an efficient and safe dose and dosing schedule of NKT-01 in induction of response in treatment of lupus nephritis.

DETAILED DESCRIPTION:
The purpose of this phase I/II study ia to establish that dose of NKT-01 which leads to complete response during a minimum of 6 cycles of treatment without causing WHO grade 3 leukopenia (WBC < 2x10^9/L). The patients suffered from uncontrolled lupus nephritis (LN) and took OCS (<= 1.0 mf/kf/day, a maximum dose of 80 mg/day) in addition to NKT-01. Therefore the aim of the open multi-center study is to determine an efficient and safe dose and dosing schedule of NKT-01 in induction of response in treatment of lupus nephritis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-70 years.
* A diagnosis of SLE according to the ACR criteria (at least 4/11 criteria).
* Sufficient signs to diagnose active SLE nephritis.
* Serum creatinine concentration of <= 5.0 mg/dL.
* Leucocyte counts >= 4000/uL.
* Receiving OCS (<= 1.0 mg/kg/day; a maximum dose of 80 mg/day).
* Prior treatment with cyclophosphamide, azathioprine, cyclosporin A, or any other immunosuppressive drugs.

Exclusion Criteria:

* Chronic infection of HIV, Hepatitis B, Hepatitis C.
* Acute infection including fungal, viral, bacterial or protozoal diseases.
* Liver toxicity (WHO CTC class 2 and higher). No adequate liver function (total bilirubin > 25 umol/L = 1.4 mg/dL unless explained otherwise (e.g. inherited, hemolysis), SGOT > 2.5 x N, SGPT > 2.5 x N).
* Pregnant or lactating women
* Female patients of child bearing age without safe method of contraception.
* Anemia (hemoglobin < 8.0 g/dL), leucopenia (leucocytes < 4000/uL unless attributable to SLE: leucocytes < 2000/uL), thrombocytopenia (platelets < 50000/uL).
* Neutrophils below 1000/uL.
* Hypogammaglobulinemia below 400 mg/dL of serum IgG.
* Any other condition that in the eyes of the investigator might have rendered the patient unsuitable for participation in the study. This especially includes major and active SLE organ involvement other than the kidney. Patients with SLE involvement of the central nervous system are not allowed to be included into the study.
* History of malignancy.
* Current participation in another trial or lass than 6 months since participation in a similar trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-10; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanns-Martin Lorenz, Professor, Principal Investigator — Heidelberg University
Locations (6):
- General Faculty Hospital, Prague, Czechia
- Germany (5):
  - Universitatsklinikum Charite, Berlin
  - Universitat Frankfurt, Frankfurt
  - University of Heidelberg, Heidelberg
  - University Hospital Mannheim, Heidelberg University, Mannheim
  - University of Regensburg, Regensburg

REFERENCES:
- [Derived] Lorenz HM, Schmitt WH, Tesar V, Muller-Ladner U, Tarner I, Hauser IA, Hiepe F, Alexander T, Woehling H, Nemoto K, Heinzel PA. Treatment of active lupus nephritis with the novel immunosuppressant 15-deoxyspergualin: an open-label dose escalation study. Arthritis Res Ther. 2011 Mar 1;13(2):R36. doi: 10.1186/ar3268. PMID 21356124

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 sites in Germany and Czech Republic from 2003 to 2007
Groups:
- Deoxyspergualin: SC, 0.5 mg/kg/day, consecutive 14 days administrations, 1 week rest, 9 cycles
Period: Overall Study
Arm/Group | Deoxyspergualin
Started | 21
Completed | 20
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: ITT population
Arm/Group | Deoxyspergualin
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: Years] | 31.3 [19 to 46]
Gender [Count of Participants; unit: Participants]
  Female | 17
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Complete and Partial Response Rate
Description: A four-point scale was defined: complete response (CR), partial response (PR), stable disease (SD) or treatment failure (TF). The response criteria were defined prior to the start of the study: for a CR, PR or SD prednisone had to be decreased to <= 7.5 mg/day, a higher dosage was automatically classified as TF. The presence of urinary erythrocyte or granular casts excluded CR. As the baseline activity of every patient is different, it was necessary to define baseline proteinuria (g/24 h) or kidney function (estimated glomerular filtration rate) as the reference value for the definition of response for every patient individually. The baseline was defined as the renal function and proteinuria level before the onset of the recent LN flare which qualified the patient for the study. Response was determined as the ratio of the proteinuria or kidney function at cycle 4, 6 or 9 to the baseline values of the individual patient.
Time Frame: Screening, Day 14 of Cycles 4, 6 and 9, up to 27 weeks
Population: ITT population
Measure: Number; unit: Percentage of participants
Arm/Group | Deoxyspergualin
Number analyzed (Participants) | 20
Percentage of participants | 55

2. Secondary Outcome: SELENA-SLEDAI Score
Description: The "Safety of Estrogen in Lupus Erythematosus National Assessment - systemic lupus erythematosus disease activity index' (SELENA-SLEDAI) document the current activity of SLE/LN. It contains 24 items (descriptors), which are differently weighed. The score has a total range of 0 - 105. As a maximum 105 score points can be reached meaning the worst disease activity.
Time Frame: Screening, the last day of Cycles 4, 6 and 9, up to 27 weeks
Population: ITT population
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Deoxyspergualin
Number analyzed (Participants) | 20
Score on a scale
  Screening | 16.9 [12 to 32]
  The last day of Cycle 4 | 12.9 [4 to 21]
  The last day of Cycle 6 | 13.7 [4 to 22]
  The last day of Cycle 9 | 11.7 [6 to 21]

3. Secondary Outcome: Treatment Days With Corticosteroids of <= 7.5 mg/Day
Description: Entry to the study was permitted for patients with doses of oral corticosteroids (OCS) of <= 1.0 mg/kg/day (maximum dose 80 mg/day).
  OCS dosage was maintained, decreased or increased according to the response to DSG.
  The number of days on which the OCS dose was <= 7.5 mg/day was counted in each cycle.
Time Frame: 1st and 9th Cycle
Population: ITT population
Measure: Mean (Full Range); unit: Days
Arm/Group | Deoxyspergualin
Number analyzed (Participants) | 20
Days
  1st Cycle | 2.8 [0 to 21]
  9th Cyvle | 18 [7 to 21]

ADVERSE EVENTS:
Time Frame: Throughout study period, up to 27 weeks
Arm/Group | Deoxyspergualin
Serious Adverse Events (participants affected / at risk) | 8/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deoxyspergualin (N=21)
Cyclophosphamide induced leucopenia (Blood and lymphatic system disorders) | 1 (1)
Leucopenia (Blood and lymphatic system disorders) | 1 (2)
Angina pectris (Cardiac disorders) | 1 (1)
Fever (General disorders) | 1 (2)
Herpes zoster (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Parodontitis, tooth infection, fever (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Increase in serum creatinine (renal failure) (Investigations) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Increased lupus activity with increased proteinuria and pain (Renal and urinary disorders) | 1 (1)
Lupus flare (arthritis, myalgia, skin rash) (Renal and urinary disorders) | 1 (1)
Renal failure (Severe proteinuria) (Renal and urinary disorders) | 1 (1)
Excision of an uterine myoma (Surgical and medical procedures) | 1 (1)
Hospitalization for a second cyclophosphamide pulse (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deoxyspergualin (N=21)
Urinary tract infection (Infections and infestations) | 6 (12)
Oral candidiasis (Infections and infestations) | 6 (7)
Vaginal candidiasis (Infections and infestations) | 4 (5)
Nasopharyngitis (Infections and infestations) | 4 (5)
Respiratory tract infection (Infections and infestations) | 3 (4)
Bronchitis (Infections and infestations) | 2 (4)
Pneumonia (Infections and infestations) | 3 (3)
Herpes simplex (Infections and infestations) | 2 (3)
Herpes zoster (Infections and infestations) | 2 (3)
Dental caries (Infections and infestations) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1)
Gasteroenteritis (Infections and infestations) | 1 (1)
Infected insect bite (Infections and infestations) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Sialoadentitis (Infections and infestations) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No